CLINICAL TRIAL: NCT06903611
Title: CAMOMILE-3: Phase III Randomized, Double-Masked, Safety and Efficacy Study of Topical Fibrinogen-Depleted Human Platelet Lysate Compared to Vehicle Control for the Treatment of Moderate to Severe Dry Eye
Brief Title: Phase III Study of Topical Fibrinogen-Depleted Human Platelet Lysate Compared to Placebo for Moderate to Severe Dry Eye
Acronym: CAMOMILE-3
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cambium Bio Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAM-101-003
Record Dates: First submitted 2025-03-25; First posted 2025-03-31 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-03

CONDITIONS: Dry Eye Disease; Dry Eye; Dry Eyes Chronic; Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: CAM-101 or vehicle control (per randomization), instill 1 drop in both eyes 4 times per day for 9 weeks. Open label use long term follow up: CAM-101, install 1 drop in both eyes 4 times per day for 43 weeks if the patient was on active IP during the 9 week randomized study or 52 weeks if the patient was on vehicle during the 9 week randomized study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Masked Placebo Controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1-Vehicle Control Group (Placebo Comparator): Vehicle Control Group - masked treatment with vehicle control for 9 weeks. Instill 1 drop in both eyes 4 times per day for 9 weeks.
  Interventions: Other: Vehicle Control
- 2-Active Treatment Group (Experimental): CAM-101 Active Group - masked treatment with CAM-101 for 9 weeks; Instill 1 drop in both eyes 4 times per day for 9 weeks. Open label use long term follow up: CAM-101, install 1 drop in both eyes 4 times per day for 43 weeks if the patient was on active IP during the 9 week randomized study or 52 weeks if the patient was on vehicle during the 9 week randomized study
  Interventions: Drug: CAM-101

INTERVENTIONS:
Drug: CAM-101 — fibrinogen depleted human platelet lysate
  Other Names: Elate Ocular; FD hPL
  Arms: 2-Active Treatment Group
Other: Vehicle Control — Plasmalyte-A
  Other Names: Placebo
  Arms: 1-Vehicle Control Group

SUMMARY:
Prospective, multicenter, randomized, vehicle-controlled, double-masked, study of CAM-101 topical ophthalmic solution compared to vehicle control followed by crossover to long-term follow-up open-label treatment with CAM-101 for one year.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety and efficacy of CAM-101 (FD hPL 30% v/v) topical ophthalmic solution after 9 weeks of treatment for moderate to severe dry eye disease and to evaluate the safety of CAM-101 (FD hPL 30%v/v) after 52-weeks of consecutive use

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects who at the time of consent are 18 years of age or older, if participating at a study site located in the U.S.; or 20 years of age or older if participating at a study site located in India.
2. Having a self-reported history of dry eye disease within the past 6 months.
3. NEI Corneal Fluorescein Staining Score in at least one eye at screening and at Day 0 (pre-randomization) that is ≥ 6≥ 6 (total score)as determined by the investigator.
4. Visual Analog Scale (VAS) Symptom Index-Eye Dryness/Eye Discomfort total score (pre-dose) that is ≥ 40 points at screening and at Day 0 (pre-randomization).
5. Willingness to have both the right and left eyes treated in the study.
6. Willingness to discontinue contact lenses and all current DED treatments except artificial tears.
7. Be able to demonstrate ability to use study medication bottle; this can be documented on study bottle used during washout period.
8. Female subjects must be either: (1) of non-childbearing potential; or, (2) of childbearing potential and using an acceptable method of birth control with a negative pregnancy test :

   1. Females of Non-childbearing Potential: Surgically sterilized (e.g., hysterectomy or bilateral oophorectomy) prior to screening; or, post-menopausal (i.e., no menstrual bleeding for at least 1 year prior to screening; or with a negative pregnancy test if less than 1 year post-menopausal).
   2. Females of Childbearing Potential: Must agree to use a highly effective acceptable form of birth control (e.g., established hormonal birth control, or double barrier method: intrauterine device plus condom or spermicidal gel plus condom) from 21 days prior to dosing until 7 days after dosing.
9. Providing written Informed Consent consistent with privacy language as per national regulations (e.g., HIPAA authorization) with signature obtained from the subject or legally authorized representative prior to the performance of any study related procedures (including withdrawal of prohibited medication.
10. Willingness and ability to comply with schedule for follow-up visits and postoperative evaluations.

    -

Exclusion Criteria:

* Subjects who meet any of the following exclusion criteria for one or both eyes at screening will not be enrolled in the study. Subjects who meet any of the following exclusion criteria for one or both eyes on Day 0 will not be randomized and will be withdrawn from the study as screen failures:

  1. Any abnormal lid anatomy or blinking function in either eye.
  2. Using any topical ocular treatment other than the following medications:

     a. Artificial Tears: Preservative-free artificial tears may be used as needed before and/or during the study. Whenever practicable, the same brand of artificial tears should be used throughout the study and its use documented in the patient diary throughout study participation.
  3. Previous ocular surgery of any type (including lacrimal, corneal and trauma), except:

     1. Non-refractive laser eye surgery of any type in either eye performed more than 3 months before screening is permitted.
     2. Refractive surgery in either eye performed more than 6 months before screening is permitted.
     3. Cataract surgery in either eye performed more than 3 months before screening is permitted
  4. Any ocular anomaly that, in the investigator's opinion, interferes with the ocular surface, including:

     1. Active ocular herpes simplex virus infection
     2. Recurrent corneal erosion
     3. Symptomatic epithelial basement membrane dystrophy
     4. Mucus fishing syndrome
     5. Giant papillary conjunctivitis
     6. Post-radiation keratitis
     7. Stevens-Johnson syndrome
     8. Corneal ulcer
     9. Abnormalities of the nasolacrimal drainage system
     10. Chemical injury
     11. Diagnosed significant anterior blepharitis and/or progressive pterygium
  5. Current history of ocular infection (viral, bacterial, fungal), disease or inflammation (e.g., uveitis) not associated with dry eye, unless the disorder or disease is, in the investigator's opinion:

     1. Stable for at least 3 months before the Screening Visit; and,
     2. Not likely to impact or possibly interfere with the interpretation of study results.
  6. Subjects with a current intraocular infection or with any other current eye or systemic condition (e.g., severe endothelial corneal dystrophy) that, in the investigator's opinion, would interfere with the dry eye evaluation or treatment, or for which the potential benefits of CAM-101 do not outweigh the risks.
  7. History of ocular allergy (including seasonal conjunctivitis) or chronic conjunctivitis other than that secondary to dry eye.
  8. Known hypersensitivity to the components of CAM-101 or the vehicle control (fibrinogen-depleted human platelet lysate; Plasma-Lyte A).
  9. Known hypersensitivity to one of the procedural medications (e.g., proparacaine, fluorescein) unless a suitable alternative medication is available.
  10. Inability to refrain from contact lens wear during the study, including the vehicle control run-in period.
  11. Anticipated need for temporary or permanent punctum plugs during the study. (If punctum plugs have been in place for at least 4 weeks prior to the screening visit, the plugs are allowed to remain in place during the study. ) Patients must remain symptomatic for DED post punctal plug insertion.
  12. Any ocular disease or ocular condition not stabilized within 1 month (30 days) before the screening visit.
  13. Any clinically significant systemic disease or condition that is inadequately controlled (e.g., diabetes, thyroid disease, autoimmune disease) or not stabilized within 4 weeks before the screening visit.
  14. Inability or unwillingness to discontinue use of autologous serum eye drops or platelet rich plasma eye drops during the 2-week run-in period and throughout the remainder of the study.
  15. Female subjects who are pregnant or lactating or plan to become pregnant during the course of the study.
  16. Subjects not under legal guardianship who, in the investigator's opinion, lack the mental capacity to provide written informed consent for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Corneal Fluorescein | 9 weeks
  • Decrease in dry eye severity from baseline after 9 weeks of CAM-101 treatment (Corneal Fluorescein Staining Index (CFSi) Score; significance evaluated at p<0.05 level); CFSi is a digital, objective, centesimal scoring system for measuring corneal fluorescein staining as an indicator of corneal surface integrity. The variability associated with the automated analysis of the corneal staining should be less than the subjective analysis of a two reader and an adjudicator model of subjectively assessing the corneal staining associated with the 4-point NEI scoring method. Corneal staining for each eye will be evaluated in each of the 5 segments for each eye. The evaluation will be scored from 0-3, where where Corneal Staining Score: 0 = none; 1 = mild; 2 = moderate; 3 = severe, and sum the total composite score for the 5 zones for each eye. Thus, each eye can have a score ranging from 0 to 15.
Eye Discomfort | 9 weeks
  • Improvement in Eye Discomfort after 9 weeks of CAM-101 treatment (VAS Symptom Index Eye Dryness/Eye Discomfort); significance evaluated at p<0.05 level); the VAS Eye Discomfort Score, is based on a continuous 100 point scale where 0 is no discomfort and 100 is intense discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: Neera Jagirdar, MD MPH, Study Director — Cambium Bio Limited